CLINICAL TRIAL: NCT00055562
Title: Multicenter, Randomized, Controlled, Double-Blind, Parallel-Group Study to Compare the Efficacy and Safety of Two CC-5013 Dose Regimens in Subjects With Metastatic Malignant Melanoma Whose Disease Has Progressed on Treatment With DTIC, IL-2 or IFN Based Therapy
Brief Title: Study to Compare the Efficacy and Safety of Two CC-5013 Dose Regimens in Subjects With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-5013-MEL-001; NCT00060281 (obsolete NCT alias)
Record Dates: First submitted 2003-03-05; First posted 2003-03-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Metastatic Melanoma; Metastatic Malignant Melanoma; Revimid; CC5013
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC 5013

SUMMARY:
Subjects are randomized to one of two treatment arms. All subjects are screened for eligibility within 28 days prior to randomization. The study consists of a treatment phase and a follow-up phase. Subjects will be treated in repeating 4 week cycles.

ELIGIBILITY:
* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Metastatic malignant melanoma now stage IV, relapsed or refractory to standard metastatic therapy.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of starting study drug.
* Patients with active brain disease, or newly diagnosed brain metastases, within 4 weeks prior to the start of study treatment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274
Dates: Start 2003-01; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (31):
- United States (25):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Southern California Norris Cancer Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - St. Francis Memorial Hospital, San Francisco, California
  - Outpatient Clinic, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - The Harold Lever Regional Cancer Center, Waterbury, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Lutheran General, Park Ridge, Illinois
  - Carle Clinic, Urbana, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Ctr, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Melanoma Center of St Louis, St Louis, Missouri
  - Biomedical Research Alliance of New York, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Linder Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Canada (6):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Qell Health Sciences Center, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - L'Hotel Dieu de Quebec, Québec, Quebec